CLINICAL TRIAL: NCT03572140
Title: Safety of Sofosbuvir Plus Daclatasvir in Patients With Chronic Hepatitis c Virus and Assessment of Resistance Associated Variants in Resistant and Relapsed Cases
Brief Title: Safety of Sofosbuvir ,Daclatasvir in HCV Patients and RAVS in Resistent and Relapsed Cases
Acronym: RAVs
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Rasha Maree Omar Ali, Principal investigator, Assiut University
Other Study IDs: RAVS in HCV
Record Dates: First submitted 2018-06-19; First posted 2018-06-28 (Actual); Last update posted 2018-06-29 (Actual); Status verified 2018-06

CONDITIONS: HCV
Keywords: HCV; Sofosbuvir; Safety; RAVs; Daclatasvir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — fresh blood sample at base line before treatment and another specimen after the end of treatment for resistent and relapsed cases
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group A: RAVS IN resistent cases after daclatasvir plus sofosbuvir treatment
  Interventions: Diagnostic Test: RAVS In relapsed and resistent cases
- group B: RAVS IN relapsed cases after daclatasvir plus sofosbuvir treatment
  Interventions: Diagnostic Test: RAVS In relapsed and resistent cases

INTERVENTIONS:
Diagnostic Test: RAVS In relapsed and resistent cases — assessment of RAVS in relapsed and resistant cases after sofosbuvir plus daclatasvir regimen

SUMMARY:
To identify side effects of Sofosbuvir/ Daclatasvir treatment regimen of chronic HCV GT-4 infection.

* To assess the occurrence and the prevalence of RAVs in patients with treatment failure and relapse after sofosbuvir and daclatasvir with assessment of their types .
* To examine the GT4 subtypes by phylogenetic analysis and baseline sequence variability among subtypes and their potential impact on treatment outcome and development of viral resistance in patients who received a regimen of Sofosbuvir/ Daclatasvir for treatment of chronic HCV GT-4.
* To assess the differences in patient demographics across GT4 subtypes.

DETAILED DESCRIPTION:
Hepatitis C virus (HCV) chronically infects approximately 120-130 million individuals worldwide .Mortality related to HCV infection has been estimated at approximately 300,000 deaths per year..

Direct antiviral agents (DAAs) effectively eradicate HCV and rapidly improve residual liver functions. Current HCV eradication rates have exceeded 90% in a very short time .

Hepatitis C virus genotype 4 (GT4) is genetically diverse, with 17 confirmed subtypes, and comprises approximately 13% of infections worldwide [3]. In Egypt, GT4 accounts for approximately 90% of infections, with subtype 4a predominating .

Sofosbuvir and daclatasvir are generally well tolerated with only a few adverse effects reported.

Hepatitis C virus resistant associated variants (RAVs) are seen in most patients who do not achieve sustained virological response (SVR). These resistance-associated mutations depend on the class of direct-acting antiviral drugs used and also vary between hepatitis C virus genotypes and subtypes.

Donaldson et al performed an analysis on four phase III clinical trials in search of common RAVs against sofosbuvir, discovering L159F, C316N, and V321A were associated with virological failure. Interestingly, this study also verified S282R mutation as associating with failure.

NS5A RAVs can be very common, with Y93H detected in up to 15% of the population and L31M in up to 6.3%. Other RAVs tend to also be fairly common detected in approximately 0.3%-3.5% of the population

ELIGIBILITY:
Inclusion Criteria:

* Anti HCV positive patients either chronic HCV or liver cirrhosis. • Detectable HCV RNA by quantitative polymerase chain reaction (PCR) prior to treatment

Exclusion Criteria:

* Co-infection with hepatitis B virus .
* Presence of malignancy before treatment.
* End-stage liver disease (Child score more than 9).
* Major co-morbid disease e.g heart failure

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cases will be recruited from the viral hepatitis clinic, department of tropical medicine, Alrajhi Liver hospital, Assiut University. The lab. work will be done by researchers from Medical Microbiology and Immunology department, Faculty of Medicine, Assiut University-University of Cincinnat, USA and Clinical pathology department, Assiut University.
Sampling Method: Non-Probability Sample
Enrollment: 297 (Estimated)
Dates: Start 2018-07-01 (Estimated); Primary Completion 2020-07-01 (Estimated); Study Completion 2020-08-01 (Estimated)

PRIMARY OUTCOMES:
relevance of HC RAVs to the outcomes of therapy with Sofosbuvir in treatment of egyptian patients infected with HCV genotype 4 | baseline
  that may be used in the future to predict the response to Sofosbuvir and this will save a huge cost for Egypt .

CONTACTS AND LOCATIONS:
Overall Officials: Ahlam Farghaly, Professor, Principal Investigator — Assiut University; haidi ramadan, Lecturer, Principal Investigator — Assiut University

REFERENCES:
- [Background] Ben Ari Z. [Chronic hepatitis C infection--eradication of the virus]. Harefuah. 2014 Jul;153(7):392-3, 433. Hebrew. PMID 25189028
- [Background] Conti F, Buonfiglioli F, Scuteri A, Crespi C, Bolondi L, Caraceni P, Foschi FG, Lenzi M, Mazzella G, Verucchi G, Andreone P, Brillanti S. Early occurrence and recurrence of hepatocellular carcinoma in HCV-related cirrhosis treated with direct-acting antivirals. J Hepatol. 2016 Oct;65(4):727-733. doi: 10.1016/j.jhep.2016.06.015. Epub 2016 Jun 24. PMID 27349488
- [Background] Reig M, Marino Z, Perello C, Inarrairaegui M, Ribeiro A, Lens S, Diaz A, Vilana R, Darnell A, Varela M, Sangro B, Calleja JL, Forns X, Bruix J. Unexpected high rate of early tumor recurrence in patients with HCV-related HCC undergoing interferon-free therapy. J Hepatol. 2016 Oct;65(4):719-726. doi: 10.1016/j.jhep.2016.04.008. Epub 2016 Apr 13. PMID 27084592
- [Background] Kamal SM, Nasser IA. Hepatitis C genotype 4: What we know and what we don't yet know. Hepatology. 2008 Apr;47(4):1371-83. doi: 10.1002/hep.22127. PMID 18240152
- [Background] Di Lello FA, Neukam K, Parra-Sanchez M, Plaza Z, Soriano V, Cifuentes C, Mira JA, Poveda E, Pineda JA. Hepatitis C virus genotype 4 in Southern and Central Spain does not originate from recent foreign migration waves. J Med Virol. 2013 Oct;85(10):1734-40. doi: 10.1002/jmv.23657. Epub 2013 Jul 16. PMID 23861220
- [Background] Donaldson EF, Harrington PR, O'Rear JJ, Naeger LK. Clinical evidence and bioinformatics characterization of potential hepatitis C virus resistance pathways for sofosbuvir. Hepatology. 2015 Jan;61(1):56-65. doi: 10.1002/hep.27375. Epub 2014 Nov 20. PMID 25123381